CLINICAL TRIAL: NCT05019729
Title: VRC 614: A Phase 1, Dose Escalation, Open-Label Clinical Trial With Experimental Controlled Human Malaria Infections (CHMI) to Evaluate Safety and Protective Efficacy of an Anti-Malaria Human Monoclonal Antibody, VRC-MALMAB0114-00-AB (L9LS), in Healthy Malaria-Naive Adults
Brief Title: Trial to Evaluate L9LS in Healthy Adults
Acronym: VRC 614
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 10000536; 000536-I
Record Dates: First submitted 2021-08-24; First posted 2021-08-25 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Malaria
Keywords: Malaria Parasitemia; Malaria Challenge; First in Human; Mosquito; Prevention
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Group 1: L9LS (1 mg/kg IV) (Experimental): L9LS (1 mg/kg) administered by intravenous (IV) infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0114-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Group 2: L9LS (5 mg/kg IV) (Experimental): L9LS (5 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0114-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Group 3: L9LS (5 mg/kg SC) (Experimental): L9LS (5 mg/kg) administered by subcutaneous (SC) injection (Day 0)
  Interventions: Drug: VRC-MALMAB0114-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Group 4: L9LS (20 mg/kg IV) (Experimental): L9LS (20 mg/kg) administered by IV infusion (Day 0)
  Interventions: Drug: VRC-MALMAB0114-00-AB; Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Group 5: CHMI Controls (Other): Control participants who did not receive L9LS and were enrolled to complete the controlled human malaria infection (CHMI)
  Interventions: Other: Plasmodium falciparum (P. falciparum) sporozoite challenge
- Group 6: L9LS (5 mg/kg IM) (Experimental): L9LS (5 mg/kg) administered by intramuscular (IM) injection (Day 0)
  Interventions: Drug: VRC-MALMAB0114-00-AB

INTERVENTIONS:
Drug: VRC-MALMAB0114-00-AB — VRC-MALMAB0114-00-AB (L9LS) is a monoclonal antibody that binds an epitope of the Plasmodium falciparum circumsporozoite protein.
  Other Names: L9LS
  Arms: Group 1: L9LS (1 mg/kg IV); Group 2: L9LS (5 mg/kg IV); Group 3: L9LS (5 mg/kg SC); Group 4: L9LS (20 mg/kg IV); Group 6: L9LS (5 mg/kg IM)
Other: Plasmodium falciparum (P. falciparum) sporozoite challenge — Participants were exposed to bites on the forearm from mosquitoes infected with Plasmodium falciparum
  Arms: Group 1: L9LS (1 mg/kg IV); Group 2: L9LS (5 mg/kg IV); Group 3: L9LS (5 mg/kg SC); Group 4: L9LS (20 mg/kg IV); Group 5: CHMI Controls

SUMMARY:
Background:

Malaria is a parasitic disease carried by mosquitoes in tropical areas. There is no vaccine to prevent malaria infection. If not treated right away, it can become serious or deadly. Researchers want to test a drug to prevent malaria.

Objective:

To test if the drug L9LS is safe and if it prevents malaria infection in people.

Eligibility:

Healthy adults ages 18-50 who have never had malaria.

Design:

Participants were screened with a medical history, physical exam, and blood tests.

Participants were divided into 6 groups:

* Three groups received L9LS by infusion into a vein, and gave blood samples before and after infusion.
* One group received L9LS injected into the fat under the skin.
* One group did not get L9LS.
* One group received L9LS injected into the muscle.

All participants who received L9LS were monitored for side effects. They had 2-3 follow-up visits during the week after the drug was given, and gave blood samples. They received a thermometer to check their temperature daily for 7 days. They received a tool to measure any redness, swelling, or bruising at the injection site.

Most participants took part in the controlled human malaria infection (CHMI) or malaria challenge to find out if L9LS prevents malaria after being bitten by infected mosquitos. Participants in the group who received L9LS injected in the muscle were enrolled after CHMI and did not take part in the CHMI. Participants who received CHMI were bitten by mosquitoes carrying the malaria parasites. A cup containing mosquitoes was placed on their arm for 5 minutes. On days 7-17 after exposure, they received daily study visits to give blood samples. Those who got malaria were treated immediately. On day 21, all CHMI participants received treatment for malaria.

Participation lasted 2-6 months, depending on study group.

DETAILED DESCRIPTION:
This was a Phase 1, open-label, dose escalation study to evaluate the safety, tolerability, pharmacokinetics and protective efficacy of an anti-malaria human monoclonal antibody, VRC-MALMAB0114-00-AB (L9LS). The primary hypothesis was that L9LS will be safe and well tolerated when administered by either intravenous (IV),subcutaneous (SC) or intramuscular (IM) routes. The secondary objectives were that L9LS will be detectable in human sera with a definable half-life and confer protection following a controlled human malaria infection (CHMI).

The study started with enrollment into Group 1. Interim safety evaluations occurred and supported continued evaluation of L9LS prior to enrolling participants into additional dose groups. All L9LS recipients in Groups 1-4 were invited to participate in the CHMI. Group 5 participants did not receive L9LS, in order to serve as the control group for the CHMI. After CHMI, all CHMI participants were evaluated for malaria parasitemia. Participants who developed blood stage infection were treated as soon as identified per protocol criteria. Participants in Group 6 received L9LS but did not take part in the CHMI.

Study follow-up continued through 24 weeks post product administration or 8 weeks post- CHMI, whichever was the most stringent.

Study Groups:

Group 1: 5 participants - 1mg/kg IV + CHMI

Group 2: 4 participants - 5 mg/kg IV + CHMI (1 participant declined to participate in the CHMI)

Group 3: 5 participants - 5 mg/ kg SC + CHMI

Group 4: 4 participants - 20 mg/kg IV + CHMI

Group 5: 9 participants - CHMI Controls (No L9LS given; 3 back up participants were not needed so were terminated early and did not participate in the CHMI)

Group 6: 5 participants - 5 mg/kg IM

ELIGIBILITY:
INCLUSION CRITERIA:

A volunteer must have met all of the following criteria to be included:

1. Able and willing to complete the informed consent process
2. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process
3. Available for clinical follow-up through the last study visit
4. 18 to 50 years of age
5. In good general health without clinically significant medical history
6. Physical examination without clinically significant findings within the 56 days prior to enrollment
7. Weight <= 115 kg (except Group 5)
8. Adequate venous access if assigned to an IV group or adequate subcutaneous tissue if assigned to an SC group
9. Willing to have blood samples collected, stored indefinitely, and used for research purposes
10. Agrees to participate in a controlled human malaria infection (CHMI) and to comply with post-CHMI follow-up requirements (except Group 6)
11. Agrees to refrain from blood donation to blood banks for 3 years following participation in CHMI (except Group 6)
12. Agrees not to travel to a malaria endemic region during the entire course of study participation (except Group 6)

    Laboratory Criteria within 56 days prior to enrollment:
13. White Blood Cell (WBC) 2,500-12,000/mm^3
14. WBC differential either within institutional normal range or accompanied by the Principal Investigator (PI) or designee approval
15. Platelets = 125,000-500,000/mm^3
16. Hemoglobin within institutional normal range or accompanied by the PI or designee approval
17. Creatinine <= 1.1 x upper limit of normal (ULN)
18. Alanine aminotransferase (ALT) <=1.25 x ULN
19. Negative for HIV infection by an FDA approved method of detection

    Laboratory Criteria documented any time during screening, prior to enrollment:
20. Negative polymerase chain reaction (PCR) for malaria (except Group 6)
21. Negative sickle cell screening test (except Group 6)
22. Electrocardiogram (ECG) without clinically significant abnormalities (examples may include: pathologic Q waves, significant ST-T wave changes, left ventricular hypertrophy, any non-sinus rhythm excluding isolated premature atrial contractions, right or left bundle branch block, advanced A-V heart block). ECG abnormalities determined by a cardiologist to be clinically insignificant as related to study participation do not preclude study enrollment (except Group 6)
23. No evidence of increased cardiovascular disease risk; defined as >10% five-year risk by the non-laboratory method (except Group 6)

    Criteria Specific to Women:
24. Postmenopausal for at least 1 year, post-hysterectomy or bilateral oophorectomy, or if of childbearing potential:

    1. Negative beta-human chorionic gonadotropin (beta-HCG) pregnancy test (urine or serum) on day of enrollment, and prior to product administration and CHMI, and
    2. Agrees to use an effective means of birth control through the duration of study participation

EXCLUSION CRITERIA:

A volunteer would have been excluded if one or more of the following conditions applied:

1. Woman who is breast-feeding or planning to become pregnant during study participation
2. Previous receipt of a malaria vaccine or anti-malaria monoclonal antibody
3. History of malaria infection
4. Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis prior to enrollment that has a reasonable risk of recurrence during the study
5. Hypertension that is not well controlled
6. Receipt of any investigational study product within 28 days prior to enrollment/product administration (Note: SARS-CoV-2 vaccines approved by emergency use authorization are not exclusionary)
7. Receipt of any live attenuated vaccines within 28 days prior to enrollment/product administration
8. Receipt of any vaccine within 2 weeks prior to enrollment/product administration
9. Bleeding disorder diagnosed by a doctor (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular injections or blood draws
10. History of a splenectomy, sickle cell disease or sickle cell trait
11. History of skeeter syndrome or anaphylactic response to mosquito-bites (except Group 6)
12. Known intolerance to chloroquine phosphate, atovaquone or proguanil (except Group 6)
13. Use or planned use of any drug with antimalarial activity that would coincide with study product or CHMI (except Group 6)
14. History of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine (except Group 6)
15. Anticipated use of medications known to cause drug reactions with chloroquine or atovaquone-proguanil (Malarone) such as cimetidine, metoclopramide, antacids, and kaolin
16. History of Sjogren's Syndrome
17. History of chronic or recurrent salivary gland disorder diagnosed by a clinician (note: an isolated occurrence of parotitis, sialadenitis, sialolithiasis, or of a salivary gland tumor is not exclusionary)
18. History of therapeutic head or neck radiation
19. Any other chronic or clinically significant medical condition that in the opinion of the investigator would jeopardize the safety or rights of the volunteer, including but not limited to: diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of: drug or alcohol abuse, asthma, autoimmune disease, infectious diseases, psychiatric disorders, heart disease, or cancer

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Wu, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) is not shared because it has limited value in a small phase 1 trial of healthy volunteers. We instead report non-IPD (aggregate) data as required in ClinicalTrials.gov.

REFERENCES:
- [Background] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949
- [Background] Ishizuka AS, Lyke KE, DeZure A, Berry AA, Richie TL, Mendoza FH, Enama ME, Gordon IJ, Chang LJ, Sarwar UN, Zephir KL, Holman LA, James ER, Billingsley PF, Gunasekera A, Chakravarty S, Manoj A, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, K C N, Murshedkar T, DeCederfelt H, Plummer SH, Hendel CS, Novik L, Costner PJ, Saunders JG, Laurens MB, Plowe CV, Flynn B, Whalen WR, Todd JP, Noor J, Rao S, Sierra-Davidson K, Lynn GM, Epstein JE, Kemp MA, Fahle GA, Mikolajczak SA, Fishbaugher M, Sack BK, Kappe SH, Davidson SA, Garver LS, Bjorkstrom NK, Nason MC, Graham BS, Roederer M, Sim BK, Hoffman SL, Ledgerwood JE, Seder RA. Protection against malaria at 1 year and immune correlates following PfSPZ vaccination. Nat Med. 2016 Jun;22(6):614-23. doi: 10.1038/nm.4110. Epub 2016 May 9. PMID 27158907
- [Background] Gaudinski MR, Berkowitz NM, Idris AH, Coates EE, Holman LA, Mendoza F, Gordon IJ, Plummer SH, Trofymenko O, Hu Z, Campos Chagas A, O'Connell S, Basappa M, Douek N, Narpala SR, Barry CR, Widge AT, Hicks R, Awan SF, Wu RL, Hickman S, Wycuff D, Stein JA, Case C, Evans BP, Carlton K, Gall JG, Vazquez S, Flach B, Chen GL, Francica JR, Flynn BJ, Kisalu NK, Capparelli EV, McDermott A, Mascola JR, Ledgerwood JE, Seder RA; VRC 612 Study Team. A Monoclonal Antibody for Malaria Prevention. N Engl J Med. 2021 Aug 26;385(9):803-814. doi: 10.1056/NEJMoa2034031. Epub 2021 Aug 11. PMID 34379916
- [Background] Lyke KE, Berry AA, Mason K, Idris AH, O'Callahan M, Happe M, Strom L, Berkowitz NM, Guech M, Hu Z, Castro M, Basappa M, Wang L, Low K, Holman LA, Mendoza F, Gordon IJ, Plummer SH, Trofymenko O, Strauss KS, Joshi S, Shrestha B, Adams M, Chagas AC, Murphy JR, Stein J, Hickman S, McDougal A, Lin B, Narpala SR, Vazquez S, Serebryannyy L, McDermott A, Gaudinski MR, Capparelli EV, Coates EE, Wu RL, Ledgerwood JE, Dropulic LK, Seder RA; VRC 612 Part C Study Team. Low-dose intravenous and subcutaneous CIS43LS monoclonal antibody for protection against malaria (VRC 612 Part C): a phase 1, adaptive trial. Lancet Infect Dis. 2023 May;23(5):578-588. doi: 10.1016/S1473-3099(22)00793-9. Epub 2023 Jan 25. PMID 36708738
- [Result] Wu RL, Idris AH, Berkowitz NM, Happe M, Gaudinski MR, Buettner C, Strom L, Awan SF, Holman LA, Mendoza F, Gordon IJ, Hu Z, Campos Chagas A, Wang LT, Da Silva Pereira L, Francica JR, Kisalu NK, Flynn BJ, Shi W, Kong WP, O'Connell S, Plummer SH, Beck A, McDermott A, Narpala SR, Serebryannyy L, Castro M, Silva R, Imam M, Pittman I, Hickman SP, McDougal AJ, Lukoskie AE, Murphy JR, Gall JG, Carlton K, Morgan P, Seo E, Stein JA, Vazquez S, Telscher S, Capparelli EV, Coates EE, Mascola JR, Ledgerwood JE, Dropulic LK, Seder RA; VRC 614 Study Team. Low-Dose Subcutaneous or Intravenous Monoclonal Antibody to Prevent Malaria. N Engl J Med. 2022 Aug 4;387(5):397-407. doi: 10.1056/NEJMoa2203067. PMID 35921449
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000536-I.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy adults were recruited for the study at the NIH Clinical Center in Bethesda, Maryland, USA.
Period: Overall Study
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 5: CHMI Controls | Group 6: L9LS (5 mg/kg IM)
Started | 5 | 4 | 5 | 4 | 9 | 5
Received Product Administration | 5 | 4 | 5 | 4 | 0 | 5
Completed Controlled Human Malaria Infection (CHMI) | 5 | 3 (One Group 2 participant declined to participate in the CHMI prior to the scheduled pre-CHMI visit and therefore was not enrolled in the CHMI group.) | 5 | 4 | 6 | 0 (Group 6 participants did not participate in the CHMI.)
Completed | 5 | 4 | 5 | 4 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Back up control participants who did not receive L9LS or CHMI because they were not needed | 0 | 0 | 0 | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Population included all enrolled participants. Age represents age at enrollment day. Weight represents weight from enrollment evaluation for participants who received L9LS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 5: CHMI Controls | Group 6: L9LS (5 mg/kg IM) | Total
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 9 | 5 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] — Age represents age at initial enrollment day.
  years | 23.4 (2.7) | 25.3 (3.3) | 26.4 (9.3) | 24.3 (3.2) | 22.9 (0.9) | 34.4 (10.6) | 25.8 (6.7)
Age, Customized [Count of Participants; unit: Participants] — Age represents age at initial enrollment day.
  Participants
    21-30 years | 5 | 4 | 4 | 4 | 9 | 2 | 28
    31-40 years | 0 | 0 | 0 | 0 | 0 | 1 | 1
    41-50 years | 0 | 0 | 1 | 0 | 0 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 4 | 0 | 6 | 0 | 15
  Male | 1 | 3 | 1 | 4 | 3 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 3 | 1 | 7
  Not Hispanic or Latino | 4 | 4 | 3 | 4 | 6 | 4 | 25
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 2 | 0 | 3
  White | 3 | 4 | 3 | 3 | 5 | 5 | 23
  More than one race | 1 | 0 | 0 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1 | 0 | 2
Weight (kg) [Mean (Standard Deviation); unit: kg] — Weight was collected at enrollment day for each group that received L9LS. Therefore, the overall weight calculation does not include the Group 5 control participants. Population: Weight was not collected for Group 5 control participants in this protocol. Per protocol, weight was only collected for participants who received L9LS.
  kg
    number analyzed (Participants) | 5 | 4 | 5 | 4 | 0 | 5 | 23
    (all) | 62.6 (7.6) | 72.2 (16.4) | 59.2 (10.4) | 76.7 (2.9) |  | 82.9 (6.9) | 70.4 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Local Reactogenicity Signs and Symptoms Within 7 Days of L9LS Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Local Symptom" is the number of participants reporting any local symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after L9LS product administration, at approximately Week 1
Population: Population included all enrolled participants who received L9LS and had safety data collected via diary card (N=23). Group 5 CHMI controls did not receive L9LS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
Participants
  Pain/Tenderness: None | 2 | 3 | 3 | 4 | 4
  Pain/Tenderness: Mild | 3 | 1 | 2 | 0 | 1
  Pain/Tenderness: Moderate | 0 | 0 | 0 | 0 | 0
  Pain/Tenderness: Severe | 0 | 0 | 0 | 0 | 0
  Pruritis (Itching): None | 5 | 4 | 4 | 4 | 5
  Pruritis (Itching): Mild | 0 | 0 | 1 | 0 | 0
  Pruritis (Itching): Moderate | 0 | 0 | 0 | 0 | 0
  Pruritis (Itching): Severe | 0 | 0 | 0 | 0 | 0
  Swelling: None | 5 | 4 | 5 | 4 | 5
  Swelling: Mild | 0 | 0 | 0 | 0 | 0
  Swelling: Moderate | 0 | 0 | 0 | 0 | 0
  Swelling: Severe | 0 | 0 | 0 | 0 | 0
  Redness: None | 5 | 4 | 4 | 4 | 5
  Redness: Mild | 0 | 0 | 1 | 0 | 0
  Redness: Moderate | 0 | 0 | 0 | 0 | 0
  Redness: Severe | 0 | 0 | 0 | 0 | 0
  Bruising: None | 4 | 4 | 5 | 4 | 5
  Bruising: Mild | 0 | 0 | 0 | 0 | 0
  Bruising: Moderate | 1 | 0 | 0 | 0 | 0
  Bruising: Severe | 0 | 0 | 0 | 0 | 0
  Any Local Symptom: None | 2 | 3 | 3 | 4 | 4
  Any Local Symptom: Mild | 2 | 1 | 2 | 0 | 1
  Any Local Symptom: Moderate | 1 | 0 | 0 | 0 | 0
  Any Local Symptom: Severe | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Systemic Reactogenicity Signs and Symptoms Within 7 Days of L9LS Product Administration
Description: Participants recorded the occurrence of solicited symptoms on a diary card for 7 days after study product administration and reviewed the diary card with clinic staff at a follow up visit. Participants were counted once for each symptom at the worst severity if they indicated experiencing the symptom more than one time at any severity during the reporting period. The number reported for "Any Systemic Symptom" is the number of participants reporting any systemic symptom at the worst severity. Reactogenicity grading (Mild, Moderate, Severe) was done using the U.S. Department of Health and Human Services, National Institutes of Health, National Institute of Allergy and Infectious Diseases, Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1.
Time Frame: 7 days after L9LS product administration, at approximately Week 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
Participants
  Malaise: None | 4 | 3 | 2 | 4 | 5
  Malaise: Mild | 1 | 1 | 3 | 0 | 0
  Malaise: Moderate | 0 | 0 | 0 | 0 | 0
  Malaise: Severe | 0 | 0 | 0 | 0 | 0
  Muscle Aches: None | 5 | 4 | 5 | 4 | 5
  Muscle Aches: Mild | 0 | 0 | 0 | 0 | 0
  Muscle Aches: Moderate | 0 | 0 | 0 | 0 | 0
  Muscle Aches: Severe | 0 | 0 | 0 | 0 | 0
  Headache: None | 4 | 3 | 3 | 4 | 4
  Headache: Mild | 1 | 1 | 1 | 0 | 1
  Headache: Moderate | 0 | 0 | 1 | 0 | 0
  Headache: Severe | 0 | 0 | 0 | 0 | 0
  Chills: None | 5 | 3 | 4 | 4 | 5
  Chills: Mild | 0 | 1 | 1 | 0 | 0
  Chills: Moderate | 0 | 0 | 0 | 0 | 0
  Chills: Severe | 0 | 0 | 0 | 0 | 0
  Nausea: None | 5 | 4 | 3 | 4 | 5
  Nausea: Mild | 0 | 0 | 1 | 0 | 0
  Nausea: Moderate | 0 | 0 | 1 | 0 | 0
  Nausea: Severe | 0 | 0 | 0 | 0 | 0
  Joint Pain: None | 5 | 3 | 5 | 4 | 5
  Joint Pain: Mild | 0 | 1 | 0 | 0 | 0
  Joint Pain: Moderate | 0 | 0 | 0 | 0 | 0
  Joint Pain: Severe | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): None | 5 | 4 | 5 | 4 | 5
  Temperature (Fever): Mild | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Moderate | 0 | 0 | 0 | 0 | 0
  Temperature (Fever): Severe | 0 | 0 | 0 | 0 | 0
  Any Systemic Symptom: None | 4 | 3 | 2 | 4 | 4
  Any Systemic Symptom: Mild | 1 | 1 | 2 | 0 | 1
  Any Systemic Symptom: Moderate | 0 | 0 | 1 | 0 | 0
  Any Systemic Symptom: Severe | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following L9LS Product Administration
Description: Unsolicited adverse event (AE) data collection included AEs of all severities from the date of product administration through the Day 28 post-product administration visit. At other time periods between study product administration and when greater than 4 weeks after the study product administration, only serious AEs (SAEs reported as a separate outcome and in the AE module) and new chronic medical conditions that required ongoing medical management (reported as a separate outcome) were recorded through the last study visit. The relationship between an AE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after L9LS product administration
Population: Population included all enrolled participants who received L9LS and had safety data collected via clinical assessment and/or lab results (N=23). Group 5 CHMI controls did not receive L9LS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
Participants
  Related to Study Product | 1 | 0 | 0 | 0 | 0
  Unrelated to Study Product | 1 | 1 | 1 | 0 | 1
  Total Number of Participants who had One or More Non-Serious Unsolicited AE after L9LS | 2 | 1 | 1 | 0 | 1

4. Primary Outcome: Number of Participants With One or More Unsolicited Non-Serious Adverse Events (AEs) Following Controlled Human Malaria Infection (CHMI)
Description: Unsolicited adverse event (AE) data collection included AEs of all severities from CHMI through the Day 28 post-CHMI visit. The relationship between an AE and CHMI was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 through 4 weeks after CHMI
Population: Population included all participants who completed CHMI (N=23). One Group 2 participant declined to participate in the CHMI prior to the scheduled pre-CHMI visit and therefore was not enrolled in the CHMI group. Group 6 L9LS (5mg/kg IM) participants did not participate in the CHMI.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 5: CHMI Controls
Number analyzed (Participants) | 5 | 3 | 5 | 4 | 6
Participants
  Related to CHMI | 0 | 0 | 0 | 0 | 0
  Unrelated to CHMI | 1 | 2 | 3 | 0 | 1
  Total Number of Participants who had One or More Non-Serious Unsolicited AE after CHMI | 1 | 2 | 3 | 0 | 1

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following L9LS Product Administration
Description: SAEs were recorded from receipt of first study product administration through the last expected study visit at Week 24. The relationship between a SAE and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after L9LS product administration through the study participation, up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With New Chronic Medical Conditions Following L9LS Product Administration
Description: New chronic medical conditions that required ongoing medical management were recorded from receipt of first study product administration through the last expected study visit at Week 24. The relationship between a new chronic medical condition and the study product was assessed by the investigator based on clinical judgment and the definitions outlined in the protocol. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Time Frame: Day 0 after L9LS product administration through the study participation, up to Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
Participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Abnormal Laboratory Measures of Safety Following L9LS Product Administration
Description: Abnormal laboratory results recorded as unsolicited adverse events (AEs) are summarized. Safety lab parameters included hematology (hemoglobin, hematocrit, mean corpuscular volume (MCV), platelets, and white blood cell (WBC), red blood cell (RBC), neutrophil, lymphocyte, monocyte, eosinophil and basophil counts) and chemistry (Comprehensive Metabolic Panel (CMP) including alanine aminotransferase (ALT) and creatinine). Complete Blood Count (CBC) with differential, CMP and ALT and creatinine results were collected at different timepoints throughout the study per the protocol's schedule of evaluations. Institutional laboratory normal ranges as well as the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1 were used.
Time Frame: Day 0 through 4 weeks after L9LS product administration
Population: Population included all enrolled participants who received L9LS and had safety data collected via laboratory results (N=23).
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
Participants
  Alanine Aminotransferase (ALT) | 0 | 0 | 0 | 0 | 1
  Creatinine | 1 | 0 | 0 | 0 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Related to Study Product | 0 | 0 | 0 | 0 | 0
  Number of Participants with one or more Abnormal Laboratory Results AE Unrelated to Study Product | 1 | 0 | 0 | 0 | 1
  Total Number of Participants who had Any Abnormal Laboratory Results Reported as AEs | 1 | 0 | 0 | 0 | 1

8. Secondary Outcome: Number of Participants Who Developed Plasmodium Falciparum (P. Falciparum) Parasitemia Following Controlled Human Malaria Infection (CHMI) Challenge
Description: Parasitemia as determined by polymerase chain reaction (PCR) up to day 21 following CHMI to determine whether IV or SC administration of L9LS mediates protection against infectious P. falciparum following CHMI
Time Frame: Up to 21 days after CHMI
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 5: CHMI Controls
Number analyzed (Participants) | 5 | 3 | 5 | 4 | 6
Participants | 1 | 0 | 1 | 0 | 6

9. Secondary Outcome: Pharmacokinetic (PK) Parameters of L9LS: Maximum Observed Serum Concentration (Cmax)
Description: Serum concentrations of L9LS by dose group following a single administration. Cmax is the peak serum concentration that L9LS achieves after it has been administered; it is determined as a maximum value on the summary pharmacokinetic (PK) curve for each study group.
Time Frame: Baseline through 24 weeks after L9LS product administration
Population: Population included all participants who received L9LS (N=23).
Measure: Mean (Standard Deviation); unit: μg/ml
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
μg/ml | 41.5 (4.7) | 164.9 (31.1) | 66.5 (3.3) | 914.2 (146.5) | 68.9 (22.3)

10. Secondary Outcome: Pharmacokinetic (PK) Parameters of L9LS: Time to Reach Maximum Observed Serum Concentration (Tmax)
Description: Tmax is the time it takes to reach Cmax of L9LS after it has been administered; it is determined based on the summary PK curve for each dose group.
Time Frame: Baseline through 24 weeks after L9LS product administration
Population: Population included all participants who received L9LS (N=23).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
days | 0.08 (0.06) | 0.06 (0.06) | 9.94 (4.06) | 0.08 (0.04) | 5.86 (2.20)

11. Secondary Outcome: Pharmacokinetic (PK) Parameters of L9LS: Beta Half-life (T1/2b)
Description: Beta half-life (T1/2b) is being reported for this study. Beta half-life (T1/2b) is the time required for half of the L9LS product to be eliminated from the serum.
Time Frame: Baseline through 24 weeks after L9LS product administration
Population: Population included all participants who received L9LS (N=23).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 4 | 5 | 4 | 5
days | 62.06 (6.29) | 70.57 (8.83) | 73.39 (16.93) | 59.45 (7.38) | 66.95 (2.54)

12. Secondary Outcome: Pharmacokinetic (PK) Parameters of L9LS: Clearance (CL) Following IV Administration
Description: Rate of L9LS elimination divided by the plasma L9LS concentration; determined based on the summary pharmacokinetic (PK) curve for each IV group.
Time Frame: Baseline through 24 weeks after L9LS product administration
Population: Population included participants who received L9LS (1 mg/kg IV, 5 mg/kg IV, and 20 mg/kg IV) intravenously (N=13).
Measure: Mean (Standard Deviation); unit: ml/day
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 4: L9LS (20 mg/kg IV)
Number analyzed (Participants) | 5 | 4 | 4
ml/day | 35.38 (3.46) | 43.54 (10.51) | 40.48 (4.65)

13. Secondary Outcome: Pharmacokinetic (PK) Parameters of L9LS: Clearance (CL/F) Following SC or IM Administration
Description: Rate of L9LS elimination divided by the plasma L9LS concentration; determined based on the summary pharmacokinetic (PK) curve for each SC and IM group. Clearance following a SC or IM administration is calculated as Clearance (CL)/Bioavailability (F).
Time Frame: Baseline through 24 weeks after L9LS product administration
Population: Population included participants who received either L9LS (5 mg/kg SC and 5 mg/kg IM) subcutaneously or intramuscularly (N=10).
Measure: Mean (Standard Deviation); unit: ml/day
Arm/Group | Group 3: L9LS (5 mg/kg SC) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 5
ml/day | 45.87 (7.17) | 60.70 (4.77)

14. Secondary Outcome: Pharmacokinetic (PK) Parameters of L9LS: Volume of Distribution at Steady-State (Vss) Following IV Administration
Description: Theoretical volume that would be necessary to contain the total amount of administered drug at the same concentration as observed in plasma. It represents the degree to which a drug is distributed in body tissue rather than the plasma and calculated based in the pharmacokinetic (PK) curve for each IV group.
Time Frame: Baseline through 24 weeks after L9LS product administration
Population: Population included participants who received L9LS (1 mg/kg IV, 5 mg/kg IV, and 20 mg/kg IV) intravenously (N=13).
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 4: L9LS (20 mg/kg IV)
Number analyzed (Participants) | 5 | 4 | 4
Liters | 3.13 (0.50) | 4.43 (1.56) | 3.42 (0.59)

15. Secondary Outcome: Pharmacokinetic (PK) Parameters of L9LS: Volume of Distribution at Steady-State (Vss/F) Following SC or IM Administration
Description: Theoretical volume that would be necessary to contain the total amount of administered drug at the same concentration as observed in plasma. It represents the degree to which a drug is distributed in body tissue rather than the plasma and calculated based in the PK curve for each SC and IM group. Volume of distribution at steady-state (Vss) following a SC or IM administration is calculated as Volume of distribution at steady-state (Vss)/Bioavailability (F).
Time Frame: Baseline through 24 weeks after L9LS product administration
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Group 3: L9LS (5 mg/kg SC) | Group 6: L9LS (5 mg/kg IM)
Number analyzed (Participants) | 5 | 5
Liters | 4.70 (0.84) | 5.77 (0.48)

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data collection included AEs of all severities for the L9LS and/or CHMI recipients only. Unsolicited AEs were recorded from the date of investigational product (IP) administration through the Day 28 post-product administration visit and from CHMI through the Day 28 post-CHMI visit. After and between the indicated time periods, only serious AEs (SAEs) and new chronic medical conditions were recorded as AEs through the last expected study visit at Week 24.
Description: Solicited AEs collected through systematic assessment for L9LS recipients only and unsolicited AEs collected for L9LS and/or CHMI recipients through non-systematic assessment represent the number and percentage of participants reporting the event. A participant with multiple experiences of the same event is counted once using the event of worst severity.
Arm/Group | Group 1: L9LS (1 mg/kg IV) | Group 2: L9LS (5 mg/kg IV) | Group 3: L9LS (5 mg/kg SC) | Group 4: L9LS (20 mg/kg IV) | Group 5: CHMI Controls | Group 6: L9LS (5 mg/kg IM)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/5 | 0/4 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/5 | 0/4 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 3/4 | 5/5 | 0/4 | 1/6 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: L9LS (1 mg/kg IV) (N=5) | Group 2: L9LS (5 mg/kg IV) (N=4) | Group 3: L9LS (5 mg/kg SC) (N=5) | Group 4: L9LS (20 mg/kg IV) (N=4) | Group 5: CHMI Controls (N=6) | Group 6: L9LS (5 mg/kg IM) (N=5)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood Creatinine Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Laryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Administration site pain (General disorders) | 3 | 1 | 2 | 0 | 0 | 1
Administration site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Administration site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Administration site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 1 | 1 | 3 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 0 | 0 | 1
Chills (General disorders) | 0 | 1 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT05019729/Prot_SAP_ICF_001.pdf